CLINICAL TRIAL: NCT01787877
Title: Inflammatory Biomarkers as Additional Tool to Neuroimaging in the Diagnosis and Management of Patients With Ischemic Stroke
Brief Title: Inflammatory Biomarkers as Tool in Diagnosis and Management of Patients With Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Saad Abu Saleh, Medical Sub Investigator, Ziv Hospital
Other Study IDs: 0064-12-ZIV; NCT01787890 (obsolete NCT alias)
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident, Inflammatory biomarkers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke patients reporting to the ER

SUMMARY:
Stroke represents the third commonest cause of death after heart disease and all types of cancer combined, and is the leading cause of long-term permanent disability among adults. Recombinant tissue plasminogen activator (tPA) is currently the only safe medical treatment for acute ischemic stroke but only a small fraction of patients are eligible for a thrombolysis treatment. Current guidelines on thrombolysis post stroke with tPA exclude its uses beyond 3 hours after stroke onset and when time of onset is unknown thus excluding many patients from potentially beneficial treatment.

For an appropriate triage and management of patients, it is essential to improve imaging techniques beyond a simple CT scan. Perfusion computed tomography (PCT), currently considered as an investigational technique, permits a quantitative determination of the cerebral perfusion within the brain. It helps distinguish salvageable ischemic penumbra from irreversibly infarcted core in acute stroke patients. This technique has therefore the potential to select patients who are most likely to benefit from thrombolysis with tPA, can be used to predict the benefit after thrombolysis and determine the suitability for other therapeutic interventions. In patients with a primary diagnosis of TIA, PCT would help to identify possible persistent cerebral ischemia but also provide important information for rapid instigation of prophylactic strategies.

The diagnosis and management of patients with ischemic stroke and TIA is challenging and is primarily based on clinical assessment in conjunction with neuroimaging. Development of specific molecular biomarkers as additional tools to support a clinical diagnosis, exclude common stroke mimics such as migraine or epileptic seizures, identify patients at risk of disease, and help guide patient treatment by predicting complications following t-PA treatment would be of great value.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments
2. Diagnosis of acute clinical stroke
3. Ages 18 and above inclusive
4. Both genders eligible for the study

Exclusion Criteria:

1. Intracerebral hemorrhage according to Computed Tomography (CT)
2. Clinical signs of infection on admission
3. Patients with chronic inflammatory disease
4. Hematologic disorders (anemia)
5. Malignant tumor
6. Renal or hepatic failure
7. Treatment with anti-inflammatory or corticosteroids drugs within a month before stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CVA reporting to the Hospital Emergency Room
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Relationship between inflammatory biomarkers and CVA patients | Follow-up 1 year
  To assess the levels over the time of selected inflammatory biomarkers, to determine the relationship between them after acute ischemic stroke and to evaluate their correlation with patients characteristics

SECONDARY OUTCOMES:
Identify patients at risk of recurrent stroke by identifying molecular biomarkers | Follow-up for 1 year
  To develop specific molecular biomarkers to support the clinical diagnosis, identify patients at risk of recurrent stroke and select the appropriate treatment

CONTACTS AND LOCATIONS:
Overall Officials: Saad Abu Saleh, MD, Study Director — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel